CLINICAL TRIAL: NCT01554644
Title: A Randomized, Double-Blind Exploratory Pilot Study Comparing Prontosan(TM) Versus Saline in the Cleansing of Chronic Leg Ulcers in Diabetic Patients
Brief Title: Prontosan Versus Saline in the Cleansing of Chronic Leg Ulcers in Diabetic Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: B. Braun Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPM-I-H-0910
Record Dates: First submitted 2012-03-06; First posted 2012-03-15 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Diabetic Complications
Keywords: Cleansing; Chronic Leg Ulcers; Diabetic Patients
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prontosan Solution and Gel (Active Comparator): ProntosanTM Wound Irrigation Solution (PHMB 0.1%, Betaine 0.1%) and ProntosanTM Wound Gel (PHMB 0.1%, Betaine 0.1%)
  Interventions: Device: Prontosan
- Saline Solution and Inert Gel (Placebo Comparator)
  Interventions: Device: Saline

INTERVENTIONS:
Device: Prontosan — Prontosan(TM) Wound Irrigation Solution (PHMB 0.1%, Betaine 0.1%) and Prontosan(TM) Wound Gel (PHMB 0.1%, Betaine 0.1%). Dressings will be changed and the treatment procedure will be repeated daily with 30ml/40 ml wound solution and 30 ml wound gel for a period of 12 weeks.
  Other Names: Double-blind intervetion; Active/placebo comparator unknown.
  Arms: Prontosan Solution and Gel
Device: Saline — Saline Wound Irrigation Solution and inert Wound Gel. Dressings will be changed and the treatment procedure will be repeated daily with 30ml/40 ml wound solution and 30 ml wound gel for a period of 12 weeks.
  Other Names: Double-blind intervetion; Active/placebo comparator unknown.
  Arms: Saline Solution and Inert Gel

SUMMARY:
This is a randomized controlled double blinded study involving two (2) investigational sites in the United States. All subjects (n=40) will receive either Prontosan Wound Irrigation Solution and Gel treatment or standard of care treatment (0.9% saline) and placebo gel. This is a 12-week study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female diabetic (type I or II) patients ≥ 18 years of age.
* Diabetic ulcer(s) present for ≥ 4 weeks located below the knee.
* A total surface area of ≥ 3 cm2 and ≤ 16 cm2.
* Willingness to wear an off-loading device if medically indicated (e.g., DH shoe or Walker).

Exclusion Criteria:

* Pregnant women and nursing mothers.
* Uncontrolled diabetes as defined by glucose levels >225 mg/dl.
* HbA1c ≥ 12%.
* Subjects with a wound infection.
* Subjects receiving antibiotic therapy within 14 days of enrollment.
* Subject with history of or clinical evidence of: Cardiac insufficiency (NYHA functional classification IV), angina pectoris (CCS functional classification IV), unstable pulmonary, renal, hepatic, endocrine or hematologic disease as determined by the Investigator (serum creatinine of > 3.0; transaminase or alkaline phosphatase levels equal to or greater than 5 times the upper limit) malnutrition (albumin < 2.5 g/dL).
* Peripheral arterial occlusive disease with a non-palpable pulse on both dorsal pedial and the posterior tibial artery.
* Presence of gangrene.
* Active rheumatic or collagen vascular disease (including rheumatoid arthritis, scleroderma, and systemic lupus erythematosus)
* Subjects that have been diagnosed with HBV, HVC, AIDS or are HIV positive.
* Osteomyelitis diagnosed by x-ray, bone biopsy, or other radiological procedure within 90 days prior to Screening Period.
* Active radiation therapy below the hip.
* Subject currently receiving, or has received oral or parenteral corticosteroids, immunosuppressive or cytotoxic agents within 30 days prior to Baseline Visit (Visit 1, Week 0) or is anticipated to require such agents during the course of the study.
* Current participation or participation in another investigational drug or medical device study within the last 30 days.
* Subjects who test positive for alcohol and or illicit drug use.
* Subjects who are unable to comprehend or comply with study requirements or ability to sign an informed consent.
* Subjects, who in the opinion of the Investigator would not be a suitable candidate for this study (reason for exclusion needs to be documented).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Relative (%) area wound size change versus baseline in respondents to treatment following a 12-week treatment period | Baseline and 12 weeks

SECONDARY OUTCOMES:
Change in absolute wound area dimensions | 12-week treatment period
Identification of bacteria present on wound bed at baseline and follow-up | 12-week treatment period
Relative change in bacterial load during treatment period | 12-week treatment period
Change in wound margins determined by color photography | 12-week treatment period
Number of "non-responders" as measured by wound size change (<50% relative wound size reduction | 12-week treatment period
Change of clinical wound infection during treatment period | 12-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: William Ennis, DO, Principal Investigator — University of Illinois Chicago; Gerit Mulder, DPM, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California San Diego, San Diego, California
  - University of Illinois Chicago, Chicago, Illinois